CLINICAL TRIAL: NCT00749073
Title: A Single-center, Prospective, Clinical Study to Assess the Clinical Application and Outcomes of Minimally Invasive Lumbar Decompression With the MILD™ Devices in Patients With Symptomatic Central Foraminal Lumbar Spinal Stenosis.
Brief Title: The Vertos MILD™ Preliminary Patient Evaluation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vertos Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C05NOV2007
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Results first posted 2013-04-04 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Spinal Stenosis; Lumbar Spinal Stenosis; Laminotomy; Laminectomy; Spine Surgery
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Percutaneous Lumbar Decompression procedure (Other): mild percutaneous lumbar decompression procedure
  Interventions: Device: Minimally Invasive Lumbar Decompression (MILD™)

INTERVENTIONS:
Device: Minimally Invasive Lumbar Decompression (MILD™) — The arthroscopic devices in this study are specialized surgical instruments intended to be used to perform percutaneous lumbar decompressive procedures for the treatment of various spinal conditions.
  Other Names: Vertos MILD™ Devices; MILD™ Tool Kit; Vertos MILD™ Tissue Sculpter; Vertos Bone Sculpter Rongeur

SUMMARY:
This is a single-center, open label, prospective clinical study to assess the clinical application and functional outcomes of symptomatic patients undergoing the Minimally Invasive Lumbar Decompression (MILD™) treatment for lumbar spinal stenosis. In this study, patient-reported outcomes over a 3 month period following treatment will be collected by the investigator. Periodic surveys for each study subject's pain, functional status, quality of life and physical examination will track outcomes following MILD™ treatment.

DETAILED DESCRIPTION:
The Vertos MILD™ devices are used for image-guided Minimally Invasive Lumbar Decompression, referred to as the MILD™ procedure. This percutaneous procedure is performed under fluoroscopic image guidance through a dorsal approach to the spine. Lumbar decompression is performed through the removal of tissue and bone, where indicated. All procedures are conducted in accordance with the product labeling and indications for use. A minimum of ten up to a maximum of twenty-five adult patients will be enrolled and followed for a period of up to 6 months. Patients with symptomatic lumbar spinal stenosis who meet the study enrollment criteria will be offered the MILD™ procedure as an alternative to surgery or continued standard non-surgical medical management.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic lumbar spinal stenosis (LSS) primarily caused by dorsal element hypertrophy.
2. Prior failure of conservative therapy.
3. Radiologic evidence of LSS (L3-L5), Ligamentum flavum > 2.5 mm, confirmed by pre op MRI and/or CT.
4. Central canal cross sectional area < 100mm2.
5. Anterior listhesis < 2 - 3mm.
6. Able to walk at least 10 feet unaided before being limited by pain.
7. Available to complete 12 weeks of follow-up.
8. A signed Informed Consent Form is obtained from the patient.
9. Adults ≥ 18 years of age.

Exclusion Criteria:

1. Prior surgery at intended treatment level.
2. History of recent spinal fractures with concurrent pain symptoms.
3. Disabling back or leg pain from causes other than LSS (e.g. acute compression fracture, metabolic neuropathy, or vascular claudication symptoms, etc.).
4. Significant disk protrusion or osteophyte formation.
5. Excessive facet hypertrophy.
6. Bleeding disorders and/or current use of anti coagulants.
7. Use of acetylsalicylic acid (ASA) and/or non-steroidal anti-inflammatory drug (NSAID) within 5 days of treatment.
8. Epidural steroids within prior three weeks.
9. Inability of the patient to lie prone for any reason with anesthesia support (e.g. chronic obstructive pulmonary disease (COPD), obesity, etc.).
10. Any potential wound healing pathologies that may compromise outcomes, including: diabetes, excessive smoking history, cancer, connective tissue diseases, recent spine radiation and severe COPD.
11. Dementia and/or inability to give informed consent.
12. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daryl R Fourney, MD, FRCSC, FACS, Principal Investigator — University of Saskatchewan, Royal University Hospital, Divison of Neurosurgery
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrolled between September 2008 and January 2009. Recruitment derived from patient pool of complex cases, all with confirmed presence of hypertrophic ligament, wait-listed for decompression laminectomy.
Groups:
- Mild Percutaneous Lumbar Decompression: The single group in this pilot study included ten patients treated for lumbar spinal stenosis of the central canal using the mild device kit to perform minimally invasive percutaneous decompression.
Period: Overall Study
Arm/Group | Mild Percutaneous Lumbar Decompression
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Mild Percutaneous Lumbar Decompression
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 62.9 (12.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Region of Enrollment [Number; unit: participants]
  Canada | 10

OUTCOME MEASURES:

1. Primary Outcome: Changes in Back Pain as Measured by a 10-point Visual Analog Scale (VAS).
Description: Clinical relevance established by change of two points or more on a ten point scale where zero represents no pain and ten represents worst pain imaginable. Mean change from baseline to Month 6 was reported with a positive number representing the baseline value minus the 6 month value.
Time Frame: Baseline and Six Months
Population: All available treated patients at six months post treatment. Mean change from baseline to Month 6 was reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mild Percutaneous Lumbar Decompression
Number analyzed (Participants) | 10
units on a scale | 3.3 (2.95)

2. Primary Outcome: Function as Measured Subjectively by the Oswestry Disability Index Patient Questionnaire
Description: Oswestry Disability Index (ODI) is used to measure permanent functional disability through a series of questions which characterize the disturbance of activities of daily living resulting from chronic back pain. The questionnaire is divided into 10 topics including pain intensity , personal care, lifting, walking, sitting, standing, sleeping, social life, traveling and employment/homemaking. Each topic is rated 0 (no pain or no limitation) to 5 (high pain or very limited physically). The worst possible score is 50 (100% disability) and best would be zero (0% disability), thus a higher ODI score indicates greater disability.
Time Frame: Baseline and Month 6
Population: All treated patients having six month follow-up were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mild Percutaneous Lumbar Decompression: The single group in this pilot study included ten patients treated for lumbar spinal stenosis of the central canal using the mild device kit to perform minimally invasive percutaneous decompression. The mean change and standard deviation between baseline (pretreatment) and Month 6 are reported, where a positive value represents the baseline value minus the 6 month value.
Arm/Group | Mild Percutaneous Lumbar Decompression
Number analyzed (Participants) | 10
units on a scale | 19.4 (22.73)

3. Primary Outcome: Quality of Life as Measured by the PCS Subscale of the Short-form 12 Question (SF-12) Survey.
Description: The 12-question SF-12v2 Health Survey is a validated generic measure of health status & outcomes, as opposed to one that targets a specific age, disease, or treatment group. The Physical Component Summary (PCS)takes into account the correlations among the Physical Functioning (PF), Role Physical (RP), Bodily Pain (BP), General Health (GH), and Vitality (VT)SF-12v2 Health Survey scales to show the broad impact on PCS. Norm-based scoring is used so each scale has the same mean (50 points) and the same standard deviation (10 points) as the general US population in 1998. Scores below 50 indicate a decline in health status, with lower scores representing worse health status. Minimally Important Difference (MID) is a measure of true clinical relevance of a difference, with suggested MID for the Physical Component Summary (PCS) being 2 to 3 points. Change from baseline to 6 months is presented, where a positive value represents the 6 month value minus the baseline value.
Time Frame: Baseline and Six months
Population: All available treated patients with six month follow-up.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mild Percutaneous Lumbar Decompression
Number analyzed (Participants) | 10
units on a scale | 6.14 (9.31) [4.40 to 11.74]

ADVERSE EVENTS:
Time Frame: Period of collection from enrollment through end of study (Month 6).
Arm/Group | Mild Percutaneous Lumbar Decompression
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
Small pilot series with short follow-up. Procedure experience of investigator limited. Minimal information available regarding appropriate patient selection, thus patient pool confined to complex cases wait-listed for more aggressive laminectomy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less